CLINICAL TRIAL: NCT02407704
Title: A Multi-level Life-span Characterization of Adult-depression and Effects of Medication and Exercise
Acronym: MEDEX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirk Erickson, PhD (Other)
Responsible Party: Sponsor-Investigator, Kirk Erickson, PhD, Associate Professor/Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MH090333-04; PRO13110090 (Other: University of Pittsburgh Institutional Review Board); MH090333 (Other Grant/Funding Number: NIH)
Record Dates: First submitted 2015-03-25; First posted 2015-04-03 (Estimated); Results first posted 2018-05-23 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2018-04

CONDITIONS: Depression; Depressive Disorder, Major; Depressive Disorder; Unipolar Depression; Major Depressive Disorder
Keywords: Exercise; Physical activity; GABA; Venlafaxine; fMRI; Spectroscopy; Reward system; BDNF; Sleep; Cognitive function; Biomarkers; Aerobic exercise
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder; Motor Activity | interventions — Venlafaxine Hydrochloride; Exercise; Lorazepam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aerobic Exercise + Venlafaxine XR (Experimental): Venlafaxine (Effexor) Extended-Release (XR) comes in capsule form and is taken by mouth. Target dose will be 150mg/d, with a maximum dose of 300mg/d (response dependent) for a minimum of 12 weeks.
  Exercise will include walking on a treadmill 1 hour 3 times/week for 12 weeks. Heart rate will be closely monitored during sessions. The intensity of the exercise will start at 50% of the age-based maximum for the first week and then increase and be maintained at 60-70% of the age-based maximum for the remainder of the intervention.
  Lorazepam may be used in the study for patients who either are already on this drug or who need it for sleep and/or anxiety. This will be administered in pill form (2mg or less per 24 hours).
  Interventions: Drug: Venlafaxine XR; Other: Aerobic Exercise; Drug: Lorazepam
- Venlafaxine XR Only (Active Comparator): Venlafaxine (Effexor) XR comes in capsule form and is taken by mouth. Target dose will be 150mg/d, with a maximum dose of 300mg/d (response dependent) for a minimum of 12 weeks.
  Lorazepam may be used in the study for patients who either are already on this drug or who need it for sleep and/or anxiety. This will be administered in pill form (2mg or less per 24 hours).
  Interventions: Drug: Venlafaxine XR; Drug: Lorazepam

INTERVENTIONS:
Drug: Venlafaxine XR
  Other Names: Effexor XR
Other: Aerobic Exercise
  Other Names: Physical Activity; Cardiovascular Exercise
  Arms: Aerobic Exercise + Venlafaxine XR
Drug: Lorazepam — Lorazepam may be used in the study for patients who either are already on this drug or who need it for sleep and/or anxiety. Patients taking another benzodiazepine will be asked to convert from their current benzodiazepine to an equivalent dose of Lorazepam (2mg or less in 24 hours). This will be administered in pill form.
  Other Names: Ativan

SUMMARY:
This pilot study aims to test a model that predicts that enhanced neurotransmitter gamma-aminobutyric acid (GABA) function in reward and affect-regulation central nervous system (CNS) circuits mediates the antidepressant effects of exercise. State-of-the-art magnetic resonance (MR) imaging, cognitive assessment, accelerometry, genetic, and inflammatory biomarkers will be acquired through the coordination of efforts from several established research programs at Western Psychiatric Institute and Clinic. This pilot study will be used as a platform for testing a causal/mediating role of GABA interneurons in reward processing and affect regulation in humans. This pilot study is not powered for testing a full causal model, but rather is intended to test overall feasibility of the intervention and acquisition of measures (see specific aim 1 below). This is a necessary prerequisite for designing a larger more definitive study of the model, which will be a component of a future grant application. Additionally, the data from this study will be used to test the clinical efficacy of exercise as an adjunctive treatment for late life depression (LLD; Specific Aim 2), as well as imaging, cognitive, and sleep aims (Specific Aims 3 and 4).

DETAILED DESCRIPTION:
Specific Aims:

Aim 1: Establish the infrastructure, protocol, and procedures for recruiting, screening, enrolling, and maintaining a sample of 30 adults (both younger adults and older adults) with major depression in a 12-week exercise intervention. The primary aim is to establish both feasibility and proof-of-concept on a wide range of biologically and clinically relevant outcomes.

Aim 2: Examine whether the 12-week physical activity + pharmacotherapy intervention reduces depressive symptoms in both younger and older adults above and beyond that of treatment as usual (TAU). Hypothesis 1: In both younger and older adults the antidepressant properties of pharmacotherapy will be augmented when combined with aerobic exercise such that the combined intervention will have higher rates of response and remission compared to only pharmacotherapy treatment.

Aim 3: Examine whether the 12-week combined physical activity and pharmacotherapy intervention changes the structural morphology in specific subfields of the hippocampus. Hypothesis 1: The medication intervention will increase hippocampal volume in the dentate gyrus and carbonic anhydrase I (CA1), but combining aerobic exercise with pharmacotherapy will magnify the effects of exercise. Hypothesis 2: The effect on hippocampal volume will be larger for older versus younger adults Aim 4: Explore how the combination of pharmacotherapy and exercise (compared with pharmacotherapy and TAU) influences a range of brain and behavioral outcomes, including resting state brain dynamics, MR spectroscopic measures of GABA, sleep efficiency, and cognitive performance. Hypothesis 1: Antidepressant pharmacotherapy will alter resting state networks, increase GABA levels, and improve sleep efficiency and cognitive performance - but these effects will be greater when combined with an aerobic exercise intervention. Hypothesis 2: These effects will be moderated by age such that the effects will be greater in older adults, supporting a dissociation between depression in younger and adults, and providing justification for fully powered study to explore these models and treatment-predictive biomarkers.

Depression is a significant global public health concern; it is the second leading cause of disability worldwide and is currently estimated to affect 350 million people. Antidepressant medications have shown to be more effective than placebo in treating depression. However, for 20-40% of individuals suffering from depression the pharmacotherapy has a slow or inadequate response. Thus, identifying alternative treatments for depression is a public health priority.

Background:

Physical activity is emerging as one of the most promising non-pharmaceutical treatments for depression. Greater amounts of self-reported physical activity are associated with fewer depressive symptoms in epidemiological studies and randomized interventions find that participation in physical activity enhances mood in depressed populations. A Cochrane review of 32 randomized interventions concluded that participation in physical activity is effective for reducing depressive symptoms compared to either no treatment or to a control condition. Importantly, antidepressants and physical activity may work through similar biological pathways to influence both mood and cognitive function. In fact, both antidepressants and physical activity increase levels of Brain-derived neurotrophic factor (BDNF) in serum and hippocampus, may mitigate or reverse hippocampal atrophy, influence expression and kinetics of serotonin and GABA pathways, regulate brain network connectivity, alter inflammatory pathways, and improve sleep efficiency. Our proposal aims to characterize these effects from the genetic to the behavioral and cognitive level, and isolate the effects of physical activity from those of medication.

Significance:

If effective, physical activity could become a first line of treatment for depression, which might also help reduce cognitive deficits, job productivity, and risk of other psychiatric conditions. Furthermore, although physical exercise has shown promise in reducing depressive symptoms, researchers still do not understand the biological pathways by which it works. One of the leading hypotheses of depression is that disruptions in GABA systems underlies the deficits. In contrast, improvements in GABA signaling is one of the ways in which exercise may improve brain function and reduce depressive symptoms. Along this line, investigators hope to determine the type of exercise (aerobic versus stretching and toning) that can be promoted in the future to improve brain function and reduce depressive symptoms. Demonstrating these links could be an important first step for developing more effective treatment plans for those suffering from depression.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 20-39 (recruitment complete) and 60-79 years old (open to recruitment)
2. Major depressive disorder (MDD), single or recurrent, as diagnosed by the PRIME-MD
3. MADRS ≥ 15
4. In-town and available to commute to Oakland for a 12-week period
5. Study nurse practitioner approval to participate in a 12-week moderate intense exercise intervention
6. Eligible to undergo MRI

Exclusion Criteria:

1. Inability to provide informed consent.
2. Modified Mini-Mental Score (3MS) less than 84 or dementia based upon Diagnostic and Statistical Manual of Mental Disorders 4th edition (DSM-IV) criteria including poor performance on the clinical neuropsychological battery, IQCODE, and all available clinical information.
3. Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms.
4. Abuse of or dependence on alcohol or other substances within the past three months
5. High risk for suicide [e.g., active suicidal ideation (SI) and/or current/recent intent or plan] AND unable to be managed safely in the clinical trial (e.g., unwilling to be hospitalized). Urgent psychiatric referral will be made in these cases.
6. Contraindication to venlafaxine XR as determined by study physician including history of intolerance of venlafaxine XR in the study target dosage range (venlafaxine XR at up to 300 mg/day).
7. Inability to communicate in English (i.e., interview cannot be conducted without an interpreter; subject largely unable to understand questions and cannot respond in English).
8. Non-correctable clinically significant sensory impairment (i.e., cannot hear well enough to cooperate with interview)
9. Unstable/uncontrolled medical illness, including delirium, hypertension, hyperlipidemia, or cerebrovascular or cardiovascular risk factors that are not under medical management.
10. Subjects taking psychotropic medications that cannot be safely tapered or discontinued prior to study initiation
11. If a patient failed a trial of venlafaxine (12 weeks of treatment with venlafaxine including at least 6 weeks on 300mg/day), he/she would not be eligible.
12. Other drugs that may affect the GABA system will be excluded (e.g., Kava, Valerian, Theanine, and GABA supplements).
13. The drug Linezolid (Zyvox) should be discontinued prior to study enrollment and should not be used during the study.
14. Exclusion criteria for MR scans include: cardiac pacemaker, aneurysm clip, cochlear implant, pregnancy, intrauterine device, shrapnel, history of metal fragments in the eye, neurostimulators, weight >250 lbs., tinnitus, or claustrophobia.
15. Current medical condition or treatment for a medical condition that could affect balance, gait, or contraindicate participation in moderate intensity physical activity.
16. Observed gait condition or use of walking assisted device that would contraindicate use of treadmill for exercise testing and intervention.
17. Current congestive heart failure, angina, uncontrolled arrhythmia, or other symptoms indicative of an increased acute risk for a cardiovascular event; within the previous 12 months having a myocardial infarction, coronary artery bypass grafting, or angioplasty; conditions requiring chronic anticoagulation (i.e. recent or recurrent DVT).
18. Eating disorders that would contraindicate physical activity.
19. Report exercise on more than three days per week for greater than 20 minutes per day over the past three months.
20. Report plans to relocate to a location not accessible to the study site or having employment, personal, or travel commitments that prohibit attendance to at least 80 percent of the scheduled intervention sessions and all of the scheduled assessments.

Ages: 60 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2015-03; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Erickson, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Butters MA, Young JB, Lopez O, Aizenstein HJ, Mulsant BH, Reynolds CF 3rd, DeKosky ST, Becker JT. Pathways linking late-life depression to persistent cognitive impairment and dementia. Dialogues Clin Neurosci. 2008;10(3):345-57. doi: 10.31887/DCNS.2008.10.3/mabutters. PMID 18979948
- [Background] Kohler S, Thomas AJ, Barnett NA, O'Brien JT. The pattern and course of cognitive impairment in late-life depression. Psychol Med. 2010 Apr;40(4):591-602. doi: 10.1017/S0033291709990833. Epub 2009 Aug 6. PMID 19656429
- [Background] Tedeschini E, Levkovitz Y, Iovieno N, Ameral VE, Nelson JC, Papakostas GI. Efficacy of antidepressants for late-life depression: a meta-analysis and meta-regression of placebo-controlled randomized trials. J Clin Psychiatry. 2011 Dec;72(12):1660-8. doi: 10.4088/JCP.10r06531. PMID 22244025
- [Background] Galper DI, Trivedi MH, Barlow CE, Dunn AL, Kampert JB. Inverse association between physical inactivity and mental health in men and women. Med Sci Sports Exerc. 2006 Jan;38(1):173-8. doi: 10.1249/01.mss.0000180883.32116.28. PMID 16394971
- [Background] Hassmen P, Koivula N, Uutela A. Physical exercise and psychological well-being: a population study in Finland. Prev Med. 2000 Jan;30(1):17-25. doi: 10.1006/pmed.1999.0597. PMID 10642456
- [Background] Barbour KA, Edenfield TM, Blumenthal JA. Exercise as a treatment for depression and other psychiatric disorders: a review. J Cardiopulm Rehabil Prev. 2007 Nov-Dec;27(6):359-67. doi: 10.1097/01.HCR.0000300262.69645.95. PMID 18197069
- [Background] Rimer J, Dwan K, Lawlor DA, Greig CA, McMurdo M, Morley W, Mead GE. Exercise for depression. Cochrane Database Syst Rev. 2012 Jul 11;(7):CD004366. doi: 10.1002/14651858.CD004366.pub5. PMID 22786489
- [Background] Blumenthal JA, Babyak MA, Doraiswamy PM, Watkins L, Hoffman BM, Barbour KA, Herman S, Craighead WE, Brosse AL, Waugh R, Hinderliter A, Sherwood A. Exercise and pharmacotherapy in the treatment of major depressive disorder. Psychosom Med. 2007 Sep-Oct;69(7):587-96. doi: 10.1097/PSY.0b013e318148c19a. Epub 2007 Sep 10. PMID 17846259
- [Background] Erickson KI, Miller DL, Roecklein KA. The aging hippocampus: interactions between exercise, depression, and BDNF. Neuroscientist. 2012 Feb;18(1):82-97. doi: 10.1177/1073858410397054. Epub 2011 Apr 29. PMID 21531985
- [Background] Garza AA, Ha TG, Garcia C, Chen MJ, Russo-Neustadt AA. Exercise, antidepressant treatment, and BDNF mRNA expression in the aging brain. Pharmacol Biochem Behav. 2004 Feb;77(2):209-20. doi: 10.1016/j.pbb.2003.10.020. PMID 14751447
- [Background] Blumenthal JA, Babyak MA, Moore KA, Craighead WE, Herman S, Khatri P, Waugh R, Napolitano MA, Forman LM, Appelbaum M, Doraiswamy PM, Krishnan KR. Effects of exercise training on older patients with major depression. Arch Intern Med. 1999 Oct 25;159(19):2349-56. doi: 10.1001/archinte.159.19.2349. PMID 10547175
- [Background] Mather AS, Rodriguez C, Guthrie MF, McHarg AM, Reid IC, McMurdo ME. Effects of exercise on depressive symptoms in older adults with poorly responsive depressive disorder: randomised controlled trial. Br J Psychiatry. 2002 May;180:411-5. doi: 10.1192/bjp.180.5.411. PMID 11983637
- [Background] Organization WH: Depression: A global public health concern, WHO Department of Mental Health and Substance Abuse,
- [Background] Steenland K, Karnes C, Seals R, Carnevale C, Hermida A, Levey A. Late-life depression as a risk factor for mild cognitive impairment or Alzheimer's disease in 30 US Alzheimer's disease centers. J Alzheimers Dis. 2012;31(2):265-75. doi: 10.3233/JAD-2012-111922. PMID 22543846
- [Background] Reynolds SL, Haley WE, Kozlenko N. The impact of depressive symptoms and chronic diseases on active life expectancy in older Americans. Am J Geriatr Psychiatry. 2008 May;16(5):425-32. doi: 10.1097/JGP.0b013e31816ff32e. PMID 18448853
- [Background] Bridle C, Spanjers K, Patel S, Atherton NM, Lamb SE. Effect of exercise on depression severity in older people: systematic review and meta-analysis of randomised controlled trials. Br J Psychiatry. 2012 Sep;201(3):180-5. doi: 10.1192/bjp.bp.111.095174. PMID 22945926
- [Background] Vaynman S, Ying Z, Gomez-Pinilla F. Hippocampal BDNF mediates the efficacy of exercise on synaptic plasticity and cognition. Eur J Neurosci. 2004 Nov;20(10):2580-90. doi: 10.1111/j.1460-9568.2004.03720.x. PMID 15548201
- [Background] Lebowitz BD, Pearson JL, Schneider LS, Reynolds CF 3rd, Alexopoulos GS, Bruce ML, Conwell Y, Katz IR, Meyers BS, Morrison MF, Mossey J, Niederehe G, Parmelee P. Diagnosis and treatment of depression in late life. Consensus statement update. JAMA. 1997 Oct 8;278(14):1186-90. PMID 9326481
- [Background] Pampallona S, Bollini P, Tibaldi G, Kupelnick B, Munizza C. Patient adherence in the treatment of depression. Br J Psychiatry. 2002 Feb;180:104-9. doi: 10.1192/bjp.180.2.104. PMID 11823317
- [Background] Teng EL, Chui HC. The Modified Mini-Mental State (3MS) examination. J Clin Psychiatry. 1987 Aug;48(8):314-8. PMID 3611032
- [Background] Wilkinson, GS, Robertson, GJ. WRAT4 Wide Range Achievement Test professional manual (4th ed.). Lutz, FL: Psychological Assessment Resources, 2006.
- [Background] Borkowski JG, Benton, AL, & Spreen O. Word Fluency and brain damage. Neuropsychologia 5:135-140, 1967.
- [Background] Wechsler, D. WAIS-IV administration and scoring manual. San Antonio, TX: Psychological Corporation, 2008.
- [Background] Delis DC, Kramer JH, Kaplan E, & Ober, BA. The California verbal learning test manual (2nd ed.). San Antonio, TX: The Psychological Corporation, 2000.
- [Derived] Gujral S, Aizenstein H, Reynolds CF 3rd, Butters MA, Grove G, Karp JF, Erickson KI. Exercise for Depression: A Feasibility Trial Exploring Neural Mechanisms. Am J Geriatr Psychiatry. 2019 Jun;27(6):611-616. doi: 10.1016/j.jagp.2019.01.012. Epub 2019 Jan 17. PMID 30797651

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were diagnosed using the SCID, and were excluded from participation if they did not meet criteria for Major Depressive Disorder. Participants were also excluded for presence of bipolar or psychotic disorders, alcohol/substance dependence within the past 3 months, or if they could not complete MRI.
Groups:
- Aerobic Exercise + Venlafaxine XR (60-79 Years of Age); Aerobic Exercise + Venlafaxine XR (20-39 Years of Age): Venlafaxine (Effexor) Extended-Release (XR) comes in capsule form and is taken by mouth. Target dose will be 150mg/d, with a maximum dose of 300mg/d (response dependent) for a minimum of 12 weeks.
  Exercise will include walking on a treadmill 1 hour 3 times/week for 12 weeks. The intensity of the exercise will start at 50% of the age-based maximum for the first week and then increase and be maintained at 60-70% of the age-based maximum for the remainder of the intervention.
  Lorazepam may be used in the study for patients who either are already on this drug or who need it for sleep and/or anxiety. This will be administered in pill form (2mg or less per 24 hours).
- Venlafaxine XR Only (60-79 Years of Age); Venlafaxine XR Only (20-39 Years of Age): Venlafaxine (Effexor) XR comes in capsule form and is taken by mouth. Target dose will be 150mg/d, with a maximum dose of 300mg/d (response dependent) for a minimum of 12 weeks.
  Lorazepam may be used in the study for patients who either are already on this drug or who need it for sleep and/or anxiety. This will be administered in pill form (2mg or less per 24 hours).
  Lorazepam: Lorazepam may be used in the study for patients who either are already on this drug or who need it for sleep and/or anxiety. Patients taking another benzodiazepine will be asked to convert from their current benzodiazepine to an equivalent dose of Lorazepam (2mg or less in 24 hours). This will be administered in pill form.
Period: Overall Study
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age)
Started | 2 | 3 | 5 | 5
Completed | 2 | 3 | 4 | 2
Not Completed | 0 | 0 | 1 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 2
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age) | Total
Number analyzed (Participants) | 2 | 3 | 5 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 5 | 5 | 12
  >=65 years | 1 | 2 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 3 | 3 | 10
  Male | 1 | 0 | 2 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 4 | 5 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 1 | 3 | 3 | 4 | 11
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 3 | 5 | 5 | 15
Montgomery Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Montgomery Asberg Depression Rating Scale measures depression severity. Scores can range from 0 to 60, with higher scores indicating higher levels of depression severity.
  units on a scale | 27.00 (0.71) | 24.33 (3.51) | 21.80 (5.81) | 25.60 (4.55) | 23.73 (4.23)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Remission
Description: Study completers will be classified as remitters vs. non-remitters. Remission will be defined as a MADRS score of 10 or less for at least two consecutive assessments. The MADRS will also be used to assess clinical response throughout the trial and to determine final medication dosage. At the end of week 6, those with a MADRS score greater than 10 will have the venlafaxine XR increased from 150 mg/d to a maximum of 300 mg/d.
Time Frame: Baseline, weekly for weeks 1 and 2, then biweekly for weeks 4-12
Population: 1 participant in the "Venlafaxine XR Only (20-39 Years of Age)" group was excluded from analyses as he/she discontinued the medication after week 8.
Measure: Count of Participants; unit: Participants
Groups:
- Venlafaxine XR Only (60-79 Years of Age); Venlafaxine XR Only (20-39 Years of Age): Venlafaxine (Effexor) XR comes in capsule form and is taken by mouth. Target dose will be 150mg/d, with a maximum dose of 300mg/d (response dependent) for a minimum of 12 weeks.
  Lorazepam may be used in the study for patients who either are already on this drug or who need it for sleep and/or anxiety. Patients taking another benzodiazepine will be asked to convert from their current benzodiazepine to an equivalent dose of Lorazepam (2mg or less in 24 hours). This will be administered in pill form.
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age)
Number analyzed (Participants) | 2 | 3 | 4 | 2
Participants | 0 | 2 | 4 | 2

2. Secondary Outcome: Inflammatory Biomarkers
Description: Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses.
Time Frame: Baseline and 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age)
Number analyzed (Participants) | 2 | 3 | 4 | 3
Participants | NA — Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses. | NA — Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses. | NA — Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses. | NA — Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses.

3. Secondary Outcome: Genetic Biomarkers
Description: Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses.
Time Frame: Baseline and 12 weeks
Population: Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age)
Number analyzed (Participants) | 2 | 3 | 4 | 3
Participants | NA — Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses. | NA — Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses. | NA — Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses. | NA — Blood samples were collected to assess biomarkers, but funding is not yet available to perform analyses.

4. Secondary Outcome: Physical Activity (SenseWear Physical Activity-monitoring Armband)
Description: This will be used to acquire objective information about physical activity. This armband is worn around the upper arm (left triceps) for 1 week and collects information about skin temperature, galvanic skin response, heat flux, and motion via a 3-axis accelerometer. This information is used in an algorithm to determine energy expenditure (EE). The device has a resolution of 1-minute indicating that we can acquire the above information on a minute-by-minute basis, which will allow us to determine both duration and intensity of activity during a normal week. Higher values indicate higher levels of activity.
Time Frame: Baseline and 12 weeks
Population: 1 participant in the Venlafaxine XR Only (20-39 Years of Age) group was excluded from analyses as he/she was non-compliant with the medication regimen, discontinuing the medication after Week 8.
Measure: Mean (Standard Deviation); unit: kcals
Groups:
- Venlafaxine XR Only (60-79 Years of Age); Venlafaxine XR Only (20-39 Years of Age): Venlafaxine (Effexor) XR comes in capsule form and is taken by mouth. Target dose will be 150mg/d, with a maximum dose of 300mg/d (response dependent) for a minimum of 12 weeks.
  Lorazepam may be used in the study for patients who either are already on this drug or who need it for sleep and/or anxiety. This will be administered in pill form (2mg or less per 24 hours).
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age)
Number analyzed (Participants) | 2 | 3 | 4 | 2
kcals
  Baseline Average Daily EE | 911.04 (604.31) | 201.64 (149.47) | 422.70 (694.21) | 731.06 (905.36)
  12 Week Average Daily EE | 324.03 (352.57) | 212.48 (216.95) | 694.21 (455.45) | 905.36 (596.69)

5. Secondary Outcome: Cardiovascular Fitness (Submaximal VO2)
Description: Cardiorespiratory fitness was measured via submaximal VO2 on a motorized treadmill while measuring oxygen utilization via Parvo Medics True one metabolic cart. The submaximal test followed a modified Balke protocol in which speed remained constant with the intensity being increased every two minutes via a raise of 2.0% of the incline. The speed was an agreed upon speed between participant and staff (between 2.0 and 4.0 mph). The submaximal VO2 was stopped when participant reached 85% of age predicted maximal heart rate (220 - age), rating of perceived exertion (RPE) equal to or greater than 15 for those who have blunted heart rate response due to beta block medication, or volitional termination by participant. Vital signs were monitored throughout the test and cool down period. Peak VO2 values for this cohort ranged from 14.04 to 36.48 ml/kg/min, with higher values correlated to higher fitness level.
Time Frame: Baseline and 12 weeks
Population: 1 participant in the "Venlafaxine XR Only (20-39 Years of Age)" group was excluded from analyses as he/she was non-compliant with the medication regimen, discontinuing the medication at Week 8.
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age)
Number analyzed (Participants) | 2 | 3 | 4 | 2
ml/kg/min
  Baseline Submaximal VO2 | 26.12 (6.78) | 27.73 (8.13) | 30.40 (7.61) | 24.17 (4.84)
  Week 12 Submaximal V02 | 24.23 (3.47) | 23.52 (3.20) | 33.89 (10.29) | 22.85 (0.77)

6. Secondary Outcome: Functional Magnetic Resonance Imaging (fMRI)
Description: Brain imaging conducted with a 7 Tesla scanner. Of particular interest were changes in hippocampal volume, GABA, and glutamate. The changes regarding hippocampal volumes are reported below. This measurement is reported in mm^3, with higher numbers indicating higher levels of gray matter in the hippocampal region. Volume is combined between right and left hemispheres. GABA and glutamate are not reported. The method used to obtain the data was being piloted for this study, and due to methodological challenges, the data is not considered to be accurate and therefore cannot be analyzed/shared.
Time Frame: Baseline and 12 weeks
Population: 2 participants were excluded from analyses due to lack of usable data at both time points.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age)
Number analyzed (Participants) | 2 | 2 | 3 | 3
mm^3
  Baseline Hippocampal Volume | 6703 (839) | 6579 (253) | 6192 (1022) | 5652 (902)
  Week 12 Hippocampal Volume | 6035 (1850) | 6511 (362) | 6040 (894) | 6091 (899)

7. Secondary Outcome: Neurocognitive Function (Neuropsychological Battery)
Description: The battery evaluates several cognitive domains. The Wechsler Adult Intelligence Scale, 4th ed. Digit Span subtest assesses attention and working memory. The Repeatable Battery of Neuropsychological Status (RBANS) measures Immediate and Delayed Memory, Attention, Language Abilities, and Visuospatial Functioning. Total index scores range from 40-155. The California Verbal Learning Test, 2nd Ed. (CVLT) assesses non-contextual verbal learning and memory. Z-scores are calculated for each of the constructs assessed by the CVLT. Subtests from the Deli-Kaplan Executive Function System (D-KEFS) assess aspects of executive functioning, including set-shifting (Trail Making Test Conditions 4 and 5: scaled score ranging from 0-19) and inhibition (Color-Word Interference Test Condition 3: weighted scaled score ranging from 1-19). Given that standardized scores are calculated for each of the neuropsychological measures, higher scores always indicate better cognitive functioning.
Time Frame: Baseline and 12 weeks
Population: 1 participant in the Venlafaxine XR Only (20-39 Years) group was excluded from analyses as he/she was non-compliant with the medication regimen. Another participant in the "Venlafaxine XR Only (60-79 Years of Age)" was excluded from analyses as he/she was unable to complete Week 12 testing due to physical limitations.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age)
Number analyzed (Participants) | 2 | 2 | 4 | 2
units on a scale
  Baseline RBANS Total Index Score | 77.00 (0.00) | 96.00 (19.80) | 101.00 (13.78) | 80.00 (7.07)
  Week 12 RBANS Total Index Score | 81.50 (3.54) | 100.50 (17.68) | 102.75 (19.74) | 85.50 (7.78)
  Baseline CVLT Long Delay Free Recall | 6.50 (7.78) | 10.00 (8.49) | 12.00 (4.55) | 8.50 (2.12)
  Week 12 CVLT Long Delay Free Recall | 3.00 (4.24) | 12.50 (3.54) | 13.50 (3.00) | 7.50 (2.12)
  Baseline DKEFS Trailmaking | 10.00 (0.00) | 11.00 (1.41) | 9.50 (1.29) | 4.50 (2.12)
  Week 12 DKEFS Trailmaking | 5.50 (3.54) | 10.50 (0.71) | 10.00 (1.41) | 5.50 (3.54)
  Baseline Digit Span Forward | 7.00 (1.41) | 7.50 (0.71) | 11.75 (2.22) | 10.00 (1.41)
  Week 12 Digit Span Forward | 7.00 (1.41) | 9.00 (1.41) | 12.00 (1.41) | 8.50 (2.12)
  Baseline Digit Span Backwards | 7.00 (2.83) | 7.00 (1.41) | 9.75 (1.71) | 7.00 (1.41)
  Week 12 Digit Span Backwards | 7.50 (2.12) | 8.50 (0.71) | 9.00 (1.83) | 6.50 (0.71)
  Baseline Color Word Interference Condition 3 | 9.00 (5.66) | 10.00 (1.41) | 11.25 (2.87) | 7.50 (0.71)
  Week 12 Color Word Interference Condition 3 | 7.50 (4.95) | 10.50 (0.71) | 9.75 (4.72) | 10.00 (2.83)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) | Venlafaxine XR Only (60-79 Years of Age) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) | Venlafaxine XR Only (20-39 Years of Age)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3 | 0/4 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/2 | 3/3 | 4/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aerobic Exercise + Venlafaxine XR (60-79 Years of Age) (N=2) | Venlafaxine XR Only (60-79 Years of Age) (N=3) | Aerobic Exercise + Venlafaxine XR (20-39 Years of Age) (N=4) | Venlafaxine XR Only (20-39 Years of Age) (N=4)
Dry mouth (General disorders) | 1 | 3 | 2 | 2
Drowsiness (General disorders) | 0 | 1 | 2 | 2
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 0
Blurred vision (Eye disorders) | 0 | 1 | 1 | 1
Headache (Nervous system disorders) | 0 | 2 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 2 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Increased appetite (General disorders) | 0 | 1 | 0 | 0
Decreased appetite (General disorders) | 0 | 1 | 2 | 2
Nausea/Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 1
Problems with urination (Renal and urinary disorders) | 0 | 0 | 0 | 1
Problems with Sexual Function (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0
Feeling light-headed on standing (General disorders) | 0 | 3 | 1 | 0
Feeling like the room is spinning (General disorders) | 0 | 0 | 1 | 0
Sweating (General disorders) | 0 | 2 | 3 | 2
Increased Body Temperature (General disorders) | 0 | 2 | 2 | 1
Tremor (General disorders) | 0 | 1 | 1 | 0
Disorientation (General disorders) | 0 | 1 | 0 | 0
Yawning (General disorders) | 1 | 2 | 0 | 1
Weight Gain (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Stiff Neck (General disorders) | 0 | 1 | 0 | 0
Bloatedness (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Agitation (General disorders) | 0 | 0 | 1 | 0
Jaw pain (General disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No